CLINICAL TRIAL: NCT05349942
Title: A Digital Method for Measurement of Palatal Asymmetry in Twins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, Professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MIRROR
Record Dates: First submitted 2022-02-15; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Identity, Body; Palate; Deformity
Keywords: Human identification; Palate morphology; Intraoral scanner; Digital dentistry
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Intraoral scanner (Planmeca Emerald) data acquisition, 3 scans are taken for each participant. Data will be exported from dedicated software (Planmeca, Romexis) and imported into GOM surface analysis software. Sample comparisons and sample preparation are performed here. The results are collected in excel spreadsheets and analyzed in SPSS statistical software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoral scanning and data acquisition (Experimental)
  Interventions: Device: Intraoral scanning and data acquisition

INTERVENTIONS:
Device: Intraoral scanning and data acquisition — Intraoral scanner data acquisition, 3 scans are taken for each participant. Data will be exported from dedicated software (Planmeca, Romexis) and imported into GOM surface analysis software. Sample comparisons and sample preparation are performed here. The results are collected in excel spreadsheets and analyzed in SPSS statistical software.

SUMMARY:
The aim of the study is to evaluate the digital palatal model as a possible tool of human identification.

DETAILED DESCRIPTION:
In this research, the investigators investigate the individual characteristics of the human upper and lower dentition and palate. The investigators use digital dentistry, record the data using an intraoral scanner, and store the extracted open source file format on a secure cloud-based server. Data validation is repeated annually. By comparing the initial and control digital samples, the investigators draw conclusions about the usability of the extracted information. The aim of the study is to develop a method and data storage protocol that will allow the patient data to be used years or decades later to replace or restore lost information.

ELIGIBILITY:
Inclusion Criteria:

* Monozygotic twins
* Same-sex Dizygotic twins
* Opposite-sex Dizygotic twins
* Triplets

Exclusion Criteria:

* Marfan-syndrome
* Non-twins

Ages: 17 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Deviation value between 3 human palatal scans | 30 second between data acquisition
  The deviation value will be measured in mm between three human palatal scans of the same individual by GOM Inspection software.
Deviation value among scans | 30 second between data acquisition
  The deviation value will be measured in mm between 9 comparisons of twin siblings by GOM Inspection software.
Deviation value between 2 scans | 30 second between data acquisition
  The deviation value will be measured in mm between 2 human palatal scans of the same individual by GOM Inspection software.
Deviation value between original scans and mirrored scans of the individual | 30 second between data acquisition
  The deviation value will be measured in mm between the original human palatal scans and mirrored human palatal scans of the same individual by GOM Inspection software.
Deviation value between original human palatal scans and mirrored human palatal scans of the twins | 30 second between data acquisition
  The deviation value will be measured in mm between the original human palatal scans and mirrored human palatal scans of twin siblings by GOM Inspection software.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Conservative Dentistry, Budapest, Hungary

REFERENCES:
- [Derived] Mikolicz A, Simon B, Roudgari A, Shahbazi A, Vag J. Human identification via digital palatal scans: a machine learning validation pilot study. BMC Oral Health. 2024 Nov 14;24(1):1381. doi: 10.1186/s12903-024-05162-0. PMID 39543590
- [Derived] Simon B, Mangano FG, Pal A, Simon I, Pellei D, Shahbazi A, Vag J. Palatal asymmetry assessed by intraoral scans: effects of sex, orthodontic treatment, and twinning. A retrospective cohort study. BMC Oral Health. 2023 May 18;23(1):305. doi: 10.1186/s12903-023-02993-1. PMID 37202781